CLINICAL TRIAL: NCT00470249
Title: A Phase II Study of Carboplatin in Combination With Gemcitabine as a Dose Dense Schedule in Patients With Locally Advanced or Metastatic Breast Cancer That Are Resistant to Anthracyclines & Taxanes
Brief Title: Carboplatin and Gemcitabine in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to difficulty in recruitment
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000542627; 2005-005164-83 (EudraCT Number)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; male breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: In this non-randomized prospective trial, patients with human epidermal growth factor 2 (HER-2)-negative locally advanced or metastatic breast cancer that was anthracycline- and taxane-resistant were treated with carboplatin at a dose equivalent to an area under the concentration-time curve of 4.5 mg/ml.min on day 1 and gemcitabine 1500 mg/m2 on day 2 of every 2-week cycle. The primary end point was overall response rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with (HER-2)-negative and anthracycline- and taxane-resistant (Experimental): Patients with human epidermal growth factor 2 (HER-2)-negative locally advanced or metastatic breast cancer that was anthracycline- and taxane-resistant
  Interventions: Drug: Carboplatin; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Carboplatin — At a dose equivalent to an area under the concentration-time curve of 4.5 mg/ml.min on day 1 of every 2-week cycle
Drug: Gemcitabine Hydrochloride — 1500 mg/m2 on day 2 of every 2-week cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin together with gemcitabine works in treating patients with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall response rate in patients with anthracycline- and taxane-resistant locally advanced or metastatic breast cancer treated with dose-dense carboplatin and gemcitabine hydrochloride.

Secondary

* Determine the overall toxicity of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.
* Determine the time to disease progression in patients treated with this regimen.
* Determine the duration of response in patients treated with this regimen.
* Determine the time to treatment failure in patients treated with this regimen.

OUTLINE: This is a nonrandomized, open-label study.

Patients receive carboplatin IV over 30 minutes on day 1 and gemcitabine hydrochloride IV over 150 minutes on day 2. Treatment repeats every 14 days for up to 9 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* DISEASE CHARACTERISTICS: histologically confirmed breast cancer, locally advanced or metastatic disease, recurrent or refractory disease, histological or cytological confirmation required for recurrence in a solitary site
* Must have received prior anthracycline and taxane as neoadjuvant, adjuvant, or metastatic therapy
* At least 1 measurable site of disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Palpable disease allowed, Lesions that have been irradiated in the advanced setting cannot be included as sites of measurable disease
* No nonmeasurable disease only, including the following:
* Bone lesions
* Leptomeningeal disease
* Ascites
* Pleural or pericardial effusion
* Inflammatory breast disease
* Lymphangitic pulmonary disease
* Abdominal masses that are not confirmed and followed by imaging techniques
* Cystic lesions
* No HER2-positive disease, defined as 3+ by IHC OR positive by FISH or chromogenic in situ hybridization
* Hormone receptor status not specified
* PATIENT CHARACTERISTICS:
* Male or female, Menopausal status not specified, ECOG performance status 0-1, Estimated life expectancy ≥ 12 weeks, Not pregnant or nursing, fertile patients must use effective contraception during and for 3 months after completion of study therapy
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* ALT or AST < 2.5 times upper limit of normal (ULN)
* Bilirubin normal
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.25 times ULN OR creatinine clearance > 40 mL/min
* Calcium ≤ 1.2 times ULN
* No concurrent serious medical or psychiatric illness, including any serious active infection incompatible with the study
* No other primary malignancy except carcinoma in situ of the cervix, adequately treated nonmelanomatous skin cancer, or any other malignancy previously treated ≥ 5 years ago with no evidence of recurrence
* No peripheral neuropathy ≥ grade 2
* PRIOR CONCURRENT THERAPY (See Disease Characteristics):
* Recovered from prior chemotherapy
* Prior hormonal therapy or immunotherapy allowed
* Antitumoral hormonal therapy must be discontinued prior to study entry
* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to the whole pelvis or to ≥ 25% of the bone marrow
* No prior gemcitabine hydrochloride, cisplatin, or carboplatin
* No other cytotoxic chemotherapy for 21 days before and for 14 days after completion of study therapy
* More than 30 days since prior treatment with a drug (not including study drug) that has not received regulatory approval for any indication at the time of study entry
* Bisphosphonate therapy may not be initiated or discontinued within 4 weeks of study entry
* No more than 1 prior course of chemotherapy for metastatic disease
* Prior chemotherapy in the adjuvant setting allowed
* Concurrent palliative radiotherapy to existing painful lesions (soft tissue or bone) allowed
* New bone pain requiring radiotherapy > 4 weeks after first study treatment considered disease progression
* New pain in a soft tissue lesion without other objective changes may be irradiated provided ≥ 1 other site of nonirradiated measurable disease exists
* No other concurrent anticancer treatment
* No concurrent tamoxifen citrate, aromatase inhibitors, or progestagens

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-07-15 (Actual); Primary Completion 2008-11-03 (Actual); Study Completion 2008-11-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete or partial response) | 8 months
  Assess the Overall response rate (complete or partial response)

SECONDARY OUTCOMES:
Overall toxicity as assessed by NCI CTCAE v3.0 | 8 months
  Summary Overall toxicity as assessed by NCI CTCAE v3.0
Overall survival | 8 months
  Assess Overall survival
Time to disease progression | 8 months
  Assess Time to disease progression
Duration of response | 8 months
  Assess Duration of response
Time to treatment failure | 8 months
  Assess Time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Murray, MD, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth, England
  - Southampton General Hospital, Southampton, England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Publication of the results — https://f1000research.com/articles/9-4